CLINICAL TRIAL: NCT02720380
Title: Buteyko Method for Children With Asthma: a Randomized Controlled Trial
Brief Title: Buteyko Method for Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Karla Morganna Pereira Pinto de Mendonça, Principal investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 562.554
Record Dates: First submitted 2016-03-07; First posted 2016-03-25 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Asthma; Child; Breathing Exercises
Keywords: Asthma; Physical Therapy Specialty; Breathing Exercises; Child; Clinical Trail
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko (Experimental): Children in the intervention group will perform 6 sessions (twice a week) of treatment with the Buteyko Method.
  Interventions: Other: Buteyko
- Asthma education (Active Comparator): Children assigned to the control group will receive, along with their parents, educational interventions in relation to asthma.
  Interventions: Other: Asthma education

INTERVENTIONS:
Other: Buteyko — Intervention will be held twice a week during 3 weeks.
  Arms: Buteyko
Other: Asthma education — Educational interventions in relation to asthma will be given to children assigned to the control group.
  Arms: Asthma education

SUMMARY:
This study has the aim to assess the effectiveness of the Buteyko method as an adjunct therapy in the treatment of children with asthma.

DETAILED DESCRIPTION:
Children from 7 to 12 years old with asthma diagnose will be included. Children in the intervention group will perform 6 sessions (twice a week) of treatment with the Buteyko Method. Children assigned to the control group will receive, along with their parents, educational interventions in relation to asthma. The investigators will assess quality of life by the PAQLQ (Paediatric Asthma Quality of Life Questionnaire), pulmonary function (spirometry) and the six-minute walk test. Vital signs, pulmonary auscultation and oxygen peripheral saturation will also be assessed during the tests. In addition, information will be collected on the numbers of hospitalizations, occurence of absence in school due to exacerbation of the disease, asthma symptoms and Beta2-agonists usage .

ELIGIBILITY:
Inclusion Criteria:

* Children from 7 up to 12 years old with asthma diagnose;
* Regular inhaled corticosteroids with no change in dose in the preceding 4 weeks;
* Children cannot present: other respiratory disease (such as cystic fibrosis, bronchiectasis, tuberculosis), retinal detachment, hypertensive crisis, congenital heart defect, pulmonary edema, history of lobectomy or lung segmentectomy, respiratory infections 15 days prior to the evaluations.

Exclusion Criteria:

* Children that are not able to perform some of the necessary procedures;
* Give up participating in the research and present acute symptoms of respiratory tract during the assessments.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life (questionnaire) | Baseline and three weeks later
  Quality of life will be assessed by the Pediatric Asthma Quality of Life Questionnaire (PAQLQ).

SECONDARY OUTCOMES:
Change in pulmonary function (spirometry) | Baseline and three weeks later
  Measured parameters (which will be expressed as percent predicted): FVC, FEV1, FEV1/FVC, FEF25-75%, PEF. PEF will be expressed as L/min.
Change in the Six-minute walk test distance | Baseline and three weeks later
Number of visits to the emergency room | Through study completion, an average of three weeks
Occurrence of absences in school | Through study completion, an average of three weeks
Occurrence of exacerbations | Through study completion, an average of three weeks
  Occurrence of asthma exacerbations or allergy episodes
Occurrence of Beta2-agonists usage | Through study completion, an average of three weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Norte (UFRN), Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No